CLINICAL TRIAL: NCT06946212
Title: Dexmedetomidine Versus Ketamine-midazolam Sedation in Awake Fiberoptic Intubation With Topical Anesthesia in Suspected Difficult Airway
Brief Title: Dexmedetomidine Versus Ketamine-midazolam Sedation in Awake Fiberoptic Intubation in Suspected Difficult Airway
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Salwa Samir El Sherbeny, Lecturer, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zu-IRB 10831-28/5-2023
Record Dates: First submitted 2025-04-13; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Awake Fiberoptic Intubation
Keywords: Sedation; Awake fiberoptic intubation
MeSH Terms: interventions — Dexmedetomidine; Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- dexmedetomidine group (Active Comparator): patients will receive an intravenous dose of dexmedetomidine at 1 mcg/kg over 10 min in 100 mL normal saline followed by continous infusion of dexmedetomidine at 0.2mcg/kg/h up to 0.7mcg/kg/hr till reaching Ramsay sedation score 2-3
  Interventions: Drug: Dexmedetomidine
- ketamine with midazolam Group (Active Comparator): patients will receive midazolam 0.02 mg /kg IV then 2 minutes later take ketamine 0.25 mg/kg IV and we will repeated this mixture till reaching Ramsay sedation score 2-3
  Interventions: Drug: Ketamine plus Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — In Dexmedetomidine group: patients received an intravenous dose of dexmedetomidine at 1 mcg/kg over 10 min in 100 mL normal saline followed by continous infusion of dexmedetomidine at 0.2mcg/kg/h up to 0.7mcg/kg/hr till reaching Ramsay sedation score 2-3
  Arms: dexmedetomidine group
Drug: Ketamine plus Midazolam — In Ketamine Midazolam group: patients received midazolam 0.02 mg /kg IV then 2 minutes later take ketamine 0.25 mg/kg IV and we will repeated this mixture till reaching Ramsay sedation score 2-3
  Arms: ketamine with midazolam Group

SUMMARY:
The goal of this clinical trial is to obtain the optimal patient's comfort and cooperation during awake fiberoptic intubation with prototype device. The main question it aims to answer is:

Which drug provides better sedative effect during awake fiberoptic intubation, dexmedetomidine or ketamine- midazolam combination with prototype supraglottic topical anaesthesia device?

DETAILED DESCRIPTION:
Awake fiberoptic intubation is the gold standard technique for managing patients with anticipated difficult airway. Conscious sedation and topical anesthesia is desirable, not only to make the procedure more tolerable and comfortable for the patient but also to ensure optimal intubating conditions. Ideal Topical Anesthesia and sedation regime for Awake fiberoptic intubation should provide comfort, cooperation, hemodynamic stability along with maintenance of spontaneous respiration. Several sedative agents have been assessed in previous studies) for this purpose (like benzodiazepine ,opioids ,ketamine , propofol and dexmedetomidine So it is important to know which has the best sedative effect dexmedetomidine or ketamine - midazolam combination with undisturbed respiratory function .

ELIGIBILITY:
Inclusion Criteria:

* Patient consent
* Age 21 to 60 years
* Both male and female
* ASA I and ASA II
* BMI : ((18.5 - 35 kg/ m2 )),
* Patient scheduled to undergo elective surgeries under general anesthesia.
* Patient with suspected difficult airway.

Exclusion Criteria:

* Sever chronic disease (cardiovascular, respiratory, renal and hepatic).
* Coagulopathies
* Mental retarted or psychiatric disorder.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Patient tolerance | During the procedure of awake fiberoptic intubation
  Patient tolerance assessed by independent observer by a five-point fiberoptic intubation comfort score (1 = no reaction, 2 = slight grimacing, 3 = heavy grimacing, 4 = verbal objection, 5 = defensive movement of head and hands

SECONDARY OUTCOMES:
Intubation score | During the procedure of awake fiberoptic intubation
  Intubation score was assessed by vocal cord movement (1 = open, 2 = moving, 3 = closing, 4 = closed) and coughing (1 = none, 2 = one gag or cough only, 3 = >1 gag or cough, but acceptable conditions, 4 = unacceptable conditions)

OTHER OUTCOMES:
Intubation time | from introduction of fibroscope till endotracheal tube in place confirmed.
  Intubation time: from introduction of fibroscope till endotracheal tube in place confirmed.
Mean arterial blood pressure | at five different times (baseline, 2 min after sedation, at the beginning of fiberscopy as it passes through the nostril, after advancing the ETT through the nasopharynx and 2 min after endotracheal intubation
  Mean arterial blood pressure ( MAP Measured in mmHg) which assessed at five different times (baseline, 2 min after sedation, at the beginning of fiberscopy as it passes through the nostril, after advancing the ETT through the nasopharynx and 2 min after endotracheal intubation).
Heart rate | Heart rate assessed at five different times (baseline, 2 min after sedation, at the beginning of fiberscopy as it passes through the nostril, after advancing the ETT through the nasopharynx and 2 min after endotracheal intubation
  Heart rate ( HR Measured in beat/ minute) which assessed at five different times (baseline, 2 min after sedation, at the beginning of fiberscopy as it passes through the nostril, after advancing the ETT through the nasopharynx and 2 min after endotracheal intubation).
Oxygen saturation | At five different times (baseline, 2 min after sedation, at the beginning of fiberscopy as it passes through the nostril, after advancing the ETT through the nasopharynx and 2 min after endotracheal intubation
  Oxygen saturation ( spO2 Measured in percentage) which assessed at five different times (baseline, 2 min after sedation, at the beginning of fiberscopy as it passes through the nostril, after advancing the ETT through the nasopharynx and 2 min after endotracheal intubation).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes